CLINICAL TRIAL: NCT05939310
Title: Improving Radical Resection Rates in Patients With Breast Cancer by Intraoperative Imaging Using Bevacizumab-IRDye800CW - the MARGIN-2 Study
Brief Title: Fluorescence Guided Surgery in Breast Cancer - The MARGIN-2 Study
Acronym: MARGIN-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10975
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Breast Cancer Invasive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescence guided surgery (Experimental): 10 mg bevacizumab-IRDye800CW, to intraoperatively assess possible tumour-positive margins.
  Interventions: Procedure: Fluorescence guided detection of tumor positive margins.

INTERVENTIONS:
Procedure: Fluorescence guided detection of tumor positive margins. — Intraoperative fluorescence imaging detection of tumor positive margins using the targeted tracer bevacizumab-IRDye800CW.

SUMMARY:
The goal of this clinical trial is to intraoperatively visualize tumour tissue in breast cancer patients using fluorescence imaging with the tracer bevacizumab-IRDye800CW and thereby enhance real-time clinical decision making, preventing postoperative tumour-positive margins.

ELIGIBILITY:
Inclusion Criteria:

* Patients are females with histologically proven carcinoma of the breast
* The carcinoma of the breast is a local disease with limited size (but tumor size ≥ 0.5cm) and in the multidisciplinary tumor board meeting breast conserving therapy is advised.
* Age ≥ 18 years
* Written informed consent has been obtained
* Women of childbearing potential (premenopausal women with intact reproductive organs and women less than two years after menopause) require use of effective contraception at least 3 months before administration of the tracer (if not, a negative serum pregnancy test has to be submitted), and they need to be willing to ensure that she or her partner uses effective contraception during the trial and for 3 months thereafter.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Non palpable breast tumor or prior surgery of this breast
* Received an investigational drug within 30 days prior to bevacizumab-IRDye800CW
* History of myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure or unstable angina within 6 months prior to enrollment
* Inadequately controlled hypertension with or without current antihypertensive medication
* Significant renal or hepatic impairment (grade II or higher deviations by CTCAE)
* History of allergy or infusion reactions bevacizumab or other monoclonal antibodies
* Pregnant or lactating women
* Patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Life expectancy < 12 weeks
* Preoperatively undetectable lymph nodes using SPECT-scan, requiring the use of patent blue

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Detection | 1 year
  To determine whether real-time tumor visualization using targeted fluorescent imaging during breast conserving therapy in breast cancer patients can be achieved intraoperatively and results in adequate assessment of the tumor margin.

SECONDARY OUTCOMES:
Detection ex-vivo imaging | 1 year
  To determine whether ex-vivo fluorescence imaging can adequately show tumor-positive margins in resected tissue samples.
Detection in-vivo imaging | 1 year
  To determine whether in-vivo fluorescence imaging can adequately show residual tumor in the cavity.
Radical resection rate | 1 year
  To analyze whether patients that in standard-of-care would have tumor-positive margins and needed additional treatment postoperatively, had a radical resection after biopsy using fluorescence guided surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen

IPD SHARING:
Plan to Share IPD: Undecided